CLINICAL TRIAL: NCT04475471
Title: WHF COVID-19 and Cardiovascular Disease Survey
Brief Title: WORLD HEART FEDERATION (WHF) COVID-19 and Cardiovascular Disease Survey
Acronym: WHF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Public Health Foundation of India (Other)
Collaborators: Centre for Chronic Disease Control, India (Other); University of Cape Town (Other); World Heart Federation, Geneva, Switzerland (Unknown)
Responsible Party: Principal Investigator, Dorairaj Prabhakaran, Prof, Public Health Foundation of India
Other Study IDs: RA1413
Record Dates: First submitted 2020-07-01; First posted 2020-07-17 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Cardiovascular Diseases
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A global study for a better understanding of the cardiovascular conditions that increase the risk of developing severe COVID-19, and a better characterization of cardiovascular complications in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
COVID-19 may be cardiotropic in a subset of patients. Both acute and pre-existing CVD impact outcomes unfavorably. It is possible that one common CVD treatment, medications that impact ACE-2 function, may impact outcomes either favorably or unfavorably.

However, studies so far have, perforce, been conducted with important limitations (e.g. small numbers, limited geographical representation, lack of data standardization for risk factors and outcomes, limited measurement, lack of appropriate adjustment for important confounders, and missing data). Considering the high global prevalence of CVD and its risk factors (e.g. hypertension and diabetes) and the suggested link with COVID19 it is urgent to initiate more robust studies to clarify the many issues early reports have engendered. So that investigators will conduct a global study for a better understanding of the cardiovascular conditions that increase the risk of developing severe COVID-19, and a better characterization of cardiovascular complications in hospitalized patients with COVID-19.

Given the continued increase in the COVID-19 cases worldwide, the study team launched WHF COVID-19 and CVD Extension Study to continue recruitment of the COVID-19 patients hospitalized in the selected high-income, middle-income, and low-income countries (sample size = 3300 patients). This extension study will provide valuable insights on the temporal trends in clinical characteristics of COVID-19, the specific cause of deaths such as sudden cardiac death and its relationship with COVID-19 infection, the impact of COVID-19 vaccination on the clinical outcomes at discharge and overall mortality, and anti-microbial resistance and its association with outcomes in COVID-19 patients.

Further, the study team is also conducting a WHF COVID-19 Long-term follow-up Study in a sample of 2000 patients from the WHF COVID-19 extension study that aims to determine the short- (3 month), medium- (6 month) and long-term (9-12 month) sequelae to COVID-19 including ongoing symptomatology, re-hospitalizations, mortality, impact on physical function and psycho-social consequences. The long-term sequelae of COVID-19 post hospital discharge are unknown, and the trajectories are likely to be heterogeneous across countries. This study will provide invaluable information about the intermediate to long-term effects of COVID-19 and the disease burden and economic impact of COVID-19 on patients with long term sequelae.

Sample Size:

1. WHF COVID-19 and CVD Study (primary cohort): 5200 participants
2. WHF Extension Study: 3300 participants
3. WHF Long term follow-up Study: approx. 2200 participants

ELIGIBILITY:
Inclusion Criteria:

* All adults (as locally defined) with confirmed COVID-19 infection who are hospitalized are eligible.

Exclusion Criteria:

* Patients for whom investigators are unable to obtain informed consent will be excluded.
* Patients who are unlikely to stay in the recruiting centre for 30 days (i.e. likely to be transferred)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in any hospital where COVID19 patients are hospitalized. Investigators will invite all WHF members from 100+ countries to identify at least two recruiting centres in their respective countries. Each centre should recruit between 50 and 200 consecutive patients. There is no limit in the number of sites to take part.
Sampling Method: Probability Sample
Enrollment: 5200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the patients for major adverse cardiovascular events (MACE) | Outcome will be assessed at discharge and 30-day follow-up visit from the hospital admission date.
  MACE is defined as the presence of any of the following CVD conditions: myocarditis, arrhythmia, heart failure [including Left ventricular ejection fraction], acute coronary event, as per the hospital admission and discharge records. Data will be collected at each site by local investigators and sent to the coordinating center. Only data outlined on the entry and outcome forms will be collected.
Assessment of the patients for Pulmonary outcomes including Pulmonary embolism, pneumonia, acute respiratory distress syndrome, need of intensive care - number of days in ICU or ICCU, need of ventilator] | at discharge and 30-day follow-up visits from the hospital admission date.
  Data will be collected at each site by local investigators and sent to the coordinating center. Only data outlined on the entry and outcome forms will be collected.
Assessment of the patients for Neurological Outcomes including stroke and Transient Ischemic Attack (TIA) | at discharge and 30-day follow-up visits from the hospital admission date.
  Data will be collected at each site by local investigators and sent to the coordinating center. Only data outlined on the entry and outcome forms will be collected.
All cause deaths | any time during the hospital admission and at 30-day follow-up.
  Specific causes of death to be evaluated using CRF including sudden cardiac death, death due to Myocardial infarction, Death due to heart failure, death due to stroke
Impact of COVID-19 vaccination on clinical outcomes - MACE (major adverse cardiovascular events) in COVID-19 hospitalized patients. | upto 30 days
  MACE is defined as the presence of any of the following CVD conditions: myocarditis, arrhythmia, heart failure [including Left ventricular ejection fraction], acute coronary event, as per the hospital admission and discharge records. Data will be collected at each site by local investigators and sent to the coordinating center. Only data outlined on the entry and outcome forms will be collected.
Persistence of long-COVID Symptoms at 1-month after discharge among survivors of COVID-19 hospitalizations. | 1-month after hospital discharge
  Questionnaires will be administered telephonically at 1-month after hospital discharge. Data will be collected at each site by local investigators and sent to the coordinating center.
Persistence of long-COVID Symptoms at 3-month after discharge among survivors of COVID-19 hospitalizations. | 3-month after hospital discharge
  Questionnaires will be administered telephonically at 3-month after hospital discharge. Data will be collected at each site by local investigators and sent to the coordinating center.
Persistence of long-COVID Symptoms at 6-month after discharge among survivors of COVID-19 hospitalizations. | 6-month after hospital discharge
  Questionnaires will be administered telephonically at 6-month after hospital discharge. Data will be collected at each site by local investigators and sent to the coordinating center.
Persistence of long-COVID Symptoms at 9-12-month after discharge among survivors of COVID-19 hospitalizations. | 9-12-month after hospital discharge
  Questionnaires will be administered telephonically at 9-12-month after hospital discharge. Data will be collected at each site by local investigators and sent to the coordinating center.

CONTACTS AND LOCATIONS:
Overall Officials: KAREN SILWA, MD, PhD, Principal Investigator — University of Cape Town; Pablo PEREL, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (32):
- Argentina (2):
  - Hospital de Clinicas of the University, Buenos Aires
  - Sanatorio Güemes Hospital, Buenos Aires
- Bangladesh (6):
  - Bangladesh Specialized Hospital (BSH), Dhaka
  - Dhaka Medical College Hospital (DMCH), Dhaka
  - DNCC Dedicated COVID-19 Hospital, Dhaka
  - Kurmitola General Hospital (KGH), Dhaka
  - Kuwait Bangladesh Friendship Hospital, Dhaka
  - Popular Medical College Hospital (PMCH), Dhaka
- University Clinical Center Republic of Srpska, Srpska, Bosnia and Herzegovina
- Colombia (2):
  - Clinica del Occidente, Columbia, Bogotá
  - Fundacion Valle del Lili, Cali
- Ghana (2):
  - Komfo Anokye Teaching Hospital, Kumasi
  - Kumasi South Regional Hospital, Kumasi
- India (5):
  - Dayanand medical college hospital, Ludhiana, Punjab
  - AIIMS, New Delhi, Delhi
  - Apollo Medical College, Jubilee Hills, Hyderabad, India, Hyderabad
  - Apollol Hopsital,, Hyderabad
  - AIIMS Jodhpur, Jodhpur
- Iran (2):
  - Amin Hospital, Isfahan
  - Khorshid Hospital, Isfahan
- Japan (2):
  - Kyoto Medical Center, Kyoto
  - National Hospital Organization Kyoto Medical Center, Japan, Kyoto
- CGTRH-MOMBASA, Kenya, Mombasa, Kenya
- UMMC, Kuala Lumpur, Malaysia
- ISSSTE Clinica Hospital, Guanajuato, Guanajuato City, Mexico
- Nigeria (2):
  - University College Hospital, Nigeria, Ibadan
  - Olabisi Onabanjo University Teaching Hospital (OOUTH), Sagamu
- Tabba Heart Institute, Karachi, Sindh, Pakistan
- University Hospital Sta Maria, Portugal, Lisbon, Portugal
- Groote Schuur Hospital, South Africa, Cape Town, South Africa
- Fedail Hospital, Khartoum, Sudan
- Levy Mwanawasa University Hospital, Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Below is the detail of the data to be collected from each patient enrolled in the study:
  * Patient demographics: age, sex, ethnicity, weight/height and education level
  * Clinical history: smoking status, hypertension, diabetes, obesity, heart failure, rheumatic heart disease, chagas, history of Coronary artery disease/ Percutaneous Coronary Interventions/ Coronary artery bypass graft surgery
  * Usual medication (before hospitalization)
  * Clinical characteristics at presentation: confirmed diagnosis of COVID-19, heart rate, blood pressure
  * Tests: ECG, ECHO, troponin, NT-proBNP and other biochemical markers
  * Medication received during hospitalization: cardiovascular and non-cardiovascular medications.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Two years after study completion and publication of main study results i.e., Dec 2023
Access Criteria: Two years after study completion and publication of main study results i.e., Dec 2023, and upon request from external researchers being sent to the study PIs and study steering committee for review and approval
URL: https://www.world-heart-federation.org/

REFERENCES:
- [Background] Nguyen JL, Yang W, Ito K, Matte TD, Shaman J, Kinney PL. Seasonal Influenza Infections and Cardiovascular Disease Mortality. JAMA Cardiol. 2016 Jun 1;1(3):274-81. doi: 10.1001/jamacardio.2016.0433. PMID 27438105
- [Background] Madjid M, Miller CC, Zarubaev VV, Marinich IG, Kiselev OI, Lobzin YV, Filippov AE, Casscells SW 3rd. Influenza epidemics and acute respiratory disease activity are associated with a surge in autopsy-confirmed coronary heart disease death: results from 8 years of autopsies in 34,892 subjects. Eur Heart J. 2007 May;28(10):1205-10. doi: 10.1093/eurheartj/ehm035. Epub 2007 Apr 17. PMID 17440221
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Yang J, Zheng Y, Gou X, Pu K, Chen Z, Guo Q, Ji R, Wang H, Wang Y, Zhou Y. Prevalence of comorbidities and its effects in patients infected with SARS-CoV-2: a systematic review and meta-analysis. Int J Infect Dis. 2020 May;94:91-95. doi: 10.1016/j.ijid.2020.03.017. Epub 2020 Mar 12. PMID 32173574
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Kwong JC, Schwartz KL, Campitelli MA, Chung H, Crowcroft NS, Karnauchow T, Katz K, Ko DT, McGeer AJ, McNally D, Richardson DC, Rosella LC, Simor A, Smieja M, Zahariadis G, Gubbay JB. Acute Myocardial Infarction after Laboratory-Confirmed Influenza Infection. N Engl J Med. 2018 Jan 25;378(4):345-353. doi: 10.1056/NEJMoa1702090. PMID 29365305
- [Background] Oudit GY, Kassiri Z, Jiang C, Liu PP, Poutanen SM, Penninger JM, Butany J. SARS-coronavirus modulation of myocardial ACE2 expression and inflammation in patients with SARS. Eur J Clin Invest. 2009 Jul;39(7):618-25. doi: 10.1111/j.1365-2362.2009.02153.x. Epub 2009 May 6. PMID 19453650
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400
- [Background] Yang C, Jin Z. An Acute Respiratory Infection Runs Into the Most Common Noncommunicable Epidemic-COVID-19 and Cardiovascular Diseases. JAMA Cardiol. 2020 Jul 1;5(7):743-744. doi: 10.1001/jamacardio.2020.0934. No abstract available. PMID 32211809
- [Background] Inciardi RM, Lupi L, Zaccone G, Italia L, Raffo M, Tomasoni D, Cani DS, Cerini M, Farina D, Gavazzi E, Maroldi R, Adamo M, Ammirati E, Sinagra G, Lombardi CM, Metra M. Cardiac Involvement in a Patient With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):819-824. doi: 10.1001/jamacardio.2020.1096. PMID 32219357
- [Background] Ribeiro AH, Ribeiro MH, Paixao GMM, Oliveira DM, Gomes PR, Canazart JA, Ferreira MPS, Andersson CR, Macfarlane PW, Meira W Jr, Schon TB, Ribeiro ALP. Automatic diagnosis of the 12-lead ECG using a deep neural network. Nat Commun. 2020 Apr 9;11(1):1760. doi: 10.1038/s41467-020-15432-4. PMID 32273514
- [Background] Alkmim MB, Silva CBG, Figueira RM, Santos DVV, Ribeiro LB, da Paixao MC, Marcolino MS, Paiva JC, Ribeiro AL. Brazilian National Service of Telediagnosis in Electrocardiography. Stud Health Technol Inform. 2019 Aug 21;264:1635-1636. doi: 10.3233/SHTI190571. PMID 31438267
- [Result] Thienemann F, Pinto F, Grobbee DE, Boehm M, Bazargani N, Ge J, Sliwa K. World Heart Federation Briefing on Prevention: Coronavirus Disease 2019 (COVID-19) in Low-Income Countries. Glob Heart. 2020 Apr 9;15(1):31. doi: 10.5334/gh.778. PMID 32489804
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Li B, Yang J, Zhao F, Zhi L, Wang X, Liu L, Bi Z, Zhao Y. Prevalence and impact of cardiovascular metabolic diseases on COVID-19 in China. Clin Res Cardiol. 2020 May;109(5):531-538. doi: 10.1007/s00392-020-01626-9. Epub 2020 Mar 11. PMID 32161990
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Fang L, Karakiulakis G, Roth M. Are patients with hypertension and diabetes mellitus at increased risk for COVID-19 infection? Lancet Respir Med. 2020 Apr;8(4):e21. doi: 10.1016/S2213-2600(20)30116-8. Epub 2020 Mar 11. No abstract available. PMID 32171062
- [Result] Smeeth L, Thomas SL, Hall AJ, Hubbard R, Farrington P, Vallance P. Risk of myocardial infarction and stroke after acute infection or vaccination. N Engl J Med. 2004 Dec 16;351(25):2611-8. doi: 10.1056/NEJMoa041747. PMID 15602021
- [Result] Alsahafi AJ, Cheng AC. The epidemiology of Middle East respiratory syndrome coronavirus in the Kingdom of Saudi Arabia, 2012-2015. Int J Infect Dis. 2016 Apr;45:1-4. doi: 10.1016/j.ijid.2016.02.004. Epub 2016 Feb 10. PMID 26875601
- [Result] Alhogbani T. Acute myocarditis associated with novel Middle east respiratory syndrome coronavirus. Ann Saudi Med. 2016 Jan-Feb;36(1):78-80. doi: 10.5144/0256-4947.2016.78. PMID 26922692
- [Result] Prabhakaran D, Singh K, Kondal D, Raspail L, Mohan B, Kato T, Sarrafzadegan N, Talukder SH, Akter S, Amin MR, Goma F, Gomez-Mesa J, Ntusi N, Inofomoh F, Deora S, Philippov E, Svarovskaya A, Konradi A, Puentes A, Ogah OS, Stanetic B, Issa A, Thienemann F, Juzar D, Zaidel E, Sheikh S, Ojji D, Lam CSP, Ge J, Banerjee A, Newby LK, Ribeiro ALP, Gidding S, Pinto F, Perel P, Sliwa K; WHF COVID-19 Study Collaborators. Cardiovascular Risk Factors and Clinical Outcomes among Patients Hospitalized with COVID-19: Findings from the World Heart Federation COVID-19 Study. Glob Heart. 2022 Jun 15;17(1):40. doi: 10.5334/gh.1128. eCollection 2022. PMID 35837356
- [Result] Sliwa K, Singh K, Raspail L, Ojji D, Lam CSP, Thienemann F, Ge J, Banerjee A, Newby LK, Ribeiro ALP, Gidding S, Pinto F, Perel P, Prabhakaran D. The World Heart Federation Global Study on COVID-19 and Cardiovascular Disease. Glob Heart. 2021 Apr 19;16(1):22. doi: 10.5334/gh.950. PMID 34040935
- [Result] Thienemann F, Chakafana G, Pineiro D, Pinto FJ, Perel P, Singh K, Eisele JL, Prabhakaran D, Sliwa K. WHF Position Statement on COVID Vaccination. Glob Heart. 2021 Apr 27;16(1):29. doi: 10.5334/gh.1027. PMID 34040942
- [Result] Prabhakaran D, Perel P, Roy A, Singh K, Raspail L, Faria-Neto JR, Gidding SS, Ojji D, Hakim F, Newby LK, Stepinska J, Lam CSP, Jobe M, Kraus S, Chuquiure-Valenzuela E, Pineiro D, Khaw KT, Bahiru E, Banerjee A, Narula J, Pinto FJ, Wood DA, Sliwa K. Management of Cardiovascular Disease Patients With Confirmed or Suspected COVID-19 in Limited Resource Settings. Glob Heart. 2020 Jul 1;15(1):44. doi: 10.5334/gh.823. PMID 32923338
- See also: WHO. Coronavirus disease 2019 (COVID-19) situation report-56 — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200316-sitrep-56-covid-19.%20pdf?sfvrsn=9fda7db2_6